CLINICAL TRIAL: NCT05501457
Title: Comparison of the Effects of Quadriceps and Gastrocnemius Muscle Training on Activities of Daily Living in COPD
Brief Title: The Effect of Different Muscle Training on Activities of Daily Living in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ahmet Payas, Director, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HititUApayas
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Quality of Life; Anxiety
Keywords: COPD; Pulmonary rehabilitation; Neuromuscular electrical stimulation
MeSH Terms: conditions — Anxiety Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The gastrocnemius group (Experimental): The patients in the first group (n=15) were given a pulmonary rehabilitation program and additionally 20 minutes of Neuromuscular electrical stimulation (Group 1) to the gastrocnemius muscle,
  Interventions: Device: Muscle strengthening with neuromuscular electrical stimulation
- The quadriceps femoris group (Experimental): The second group was given a pulmonary rehabilitation program and an additionally 20 minutes of neuromuscular electrical stimulation to the quadriceps femoris muscle (Group 2),
  Interventions: Device: Muscle strengthening with neuromuscular electrical stimulation
- The control group (Experimental): The third group, which was the control group, was given only a pulmonary rehabilitation program (Group 3).
  Interventions: Device: Muscle strengthening with neuromuscular electrical stimulation

INTERVENTIONS:
Device: Muscle strengthening with neuromuscular electrical stimulation — The effect of peripheral muscle strengthening training in addition to pulmonary rehabilitation in COPD patients on the patient's performance will be examined.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) contributes significantly to global morbidity and mortality; It is a disease that affects an estimated 210 million people worldwide and is the third most common cause of death. COPD is identified by persistent airflow limitation and is associated with progressively worsening lung function, dyspnea, health-related quality of life (HRQOL), and impaired exercise capacity. Poor exercise capacity is a common finding of chronic obstructive pulmonary disease (COPD). Central cardiopulmonary factors, respiratory muscle dysfunction, gas exchange abnormalities, and skeletal muscle dysfunction all play a role in limiting exercise capacity The aim of this study is to investigate the effects of neuromuscular electrical stimulation applied to different muscle groups (quadriceps femoris and gastrocnemius muscles) on exercise performance and quality of life in patients with stable COPD and compare it with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-75 years old,
* Diagnosed as group B stable COPD according to GOLD criteria by a pulmonologist,
* PaO2 >55 mm Hg, PaCO2 <45 mmHg in room air.

Exclusion Criteria:

* Exacerbation,
* Cor pulmonale or respiratory muscle fatigue (abdominal paradoxical breathing),
* Cardiac instability (with acute MI, congestive heart failure, or uncontrollable arrhythmia),
* Musculoskeletal disorder (conditions affecting exercise ability),
* Difficulty communicating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test (6 MWT): | 4 weeks
  they could walk for 6 minutes, according to heart rate, blood pressure, respiratory rate, finger oxygen saturation, the walking distance at the end of walking, and dyspnea score according to the Modified Borg Scale (MBS) at the beginning and end of walking was recorded. Change from baseline 6 Minute walking performance after 4 weeks will be examined.

SECONDARY OUTCOMES:
Modified Borg Scale (MBS): | 4 weeks
  It consists of 10 items that define the severity of dyspnea according to their degrees. Change from baseline dyspnea after 4 weeks will be examined.
St. George's Respiratory Questionnaire (SGRQ): | 4 weeks
  This questionnaire was developed specifically to determine the severity of the disease in COPD and asthma. Change from baseline severity of the disease after 4 weeks will be examined.
Beck Depression Inventory (BDI): | 4 weeks
  It measures the behavioral findings of depression in adolescents and adults. Change from baseline depression status after 4 weeks will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Payas, Dr, Study Director — HİTİT UNIVERSITY CORUM EROL OLCOK EDUCATION AND RESEARCH HOSPITAL
Locations (1):
- Hititi University Sungurlu Vocational School, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A short summary of the study can be shared.